CLINICAL TRIAL: NCT01802190
Title: Prevalence of POU4F3 (DFNA15) and SLC17A8 (DFNA25) Genes Mutations in Dominant Autosomal Deafness and Phenotypic Characterization of Carrier Patients.
Brief Title: Prevalence of POU4F3 and SLC17A8 Mutations
Status: Terminated | Type: Observational
Why Stopped: No convincing results
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8640; 2010-A00561-38 (Other: ID-RCB)
Record Dates: First submitted 2012-07-24; First posted 2013-03-01 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-04

CONDITIONS: Familial Deafness
Keywords: Genetic deafness; SLC17A8 et POU4F3 genes

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deafness patients: Deafness patients
  Interventions: Genetic: Deafness patients

INTERVENTIONS:
Genetic: Deafness patients — SLC17A8 et POU4F3 mutations genes analysis on blood samples of deafness patients.
  Other Names: SLC17A8 et POU4F3 mutations genes analysis

SUMMARY:
The study will allow to identify the prevalence of the SLC17A8 gene mutations in patients suffering from deafness. This phenotype also corresponds to DFNA15 deafness caused by POU4F3 : mutations of this gene will be screened as well.

DETAILED DESCRIPTION:
DFNA are characterized as progressive bilateral deafness. To date, 21 genes and 57 loci are involved in these dominant deafness, with an unknown prevalence.A 22nd gene responsible of the disease has been found. This SLC17A8 gene encodes for the VGLUT3 protein which is specifically expressed in sensorial cells of the audition. VGlut3-/- mice present a deep deafness due to a deficiency of neurotransmitter release, although sensorial cells and neurons are intact. This kind of deafness is an ideal candidate for a genetic therapy because of the cells integrity.Mutations of SLC17A8 gene have been found in 2 american families that suffer from progressive deafness.The study aims to look for european families from the Mediterranean basin, which carry SLC17A8 gene mutations, and may benefit in a medium-term from genetic therapy. The study will allow to identify the prevalence of the SLC17A8 gene mutations in patients suffering from deafness. This phenotype also corresponds to DFNA15 deafness caused by POU4F3 : mutations of this gene will be screened as well.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with a

  1. suggestive neurosensory Deafness: The characteristics of the deafness will be determined from the data of the questionnaire, of the interrogation, the examination and results of the tonal audiometry.

     *Neurosensory deafness: Audiometrics measurement(difference between the tonal audiometric average loss for the frequencies 0,5, 1, 2 and 4 kHz in air conduction and in osseous conduction) < 15 dB for each of both ears.
     * Bilateral symetric: difference between the audiometric thresholds of both ears < or = 15 dB for at least two frequencies.
     * Light to severe: The degree of deafness is defined according to the following classification (moderate hearing loss calculated on the frequencies 500 Hz, 1, 2 and 4 kHz): light hearing deficiency from 20 to 40 dB, moderate hearing deficiency of 40 to 70 dB, severe hearing deficiency of 70 in 90 dB and deep hearing deficiency beyond 90 dB.
     * Whose thresholds frequency by frequency in tonal audiometry (air conduction) are superior to the thresholds of the 90th percentile of the standard ISO 7029.
     * Without environmental exposition factors.
  2. Dominant autosomal transmission diagnosed from one of the following elements:

     * Deafness at a father and his son
     * Deafness at a father and his daughter outside a suggestive context of a dominant form X-related. (deep deafness at the father and light to moderate deafness in daughter)
     * Deafness at a mother and her daughter
     * Deafness at a mother and her son outside a suggestive context of a dominant X-related(light to moderate deafness at the mother, and deep deafness at the son)
     * Deafness at a patient whose a dead parent had a sure or likely deafness according to the criteria of diagnosis mentioned previously
  3. given the consent to participate at this clinical study

Exclusion Criteria:

* Suggestive symptom of a polymalformative syndrom
* familial Consanguinity
* Age < 18 years
* Deafness of transmission or mixed
* Deafness of asymmetric or fluctuating perception
* Prelingual deep Deafness
* Pathology of the ear (otospongiose, disease of Ménière, neurinome of the acoustics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Deafness patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
SLC17A8 et POU4F3 mutations genes analysis | up to 1 year
  The mutations will be screened by direct sequencing

SECONDARY OUTCOMES:
Phenotypic characterization of the carrier patients | up to 1 year
  The phenotypic characterization will be assessed by usual tests for genetic deafness (audiometry, electro-physiological explorations)

CONTACTS AND LOCATIONS:
Overall Officials: Michel MONDAIN, PU-PH, Principal Investigator — CHRU Montpellier
Locations (1):
- Mondain Michel, Montpellier, France